CLINICAL TRIAL: NCT01890720
Title: Use of Incisional Negative Pressure Wound Therapy for Prevention of Postoperative Infections Following Caesarean Section in Women With BMI >=30
Brief Title: Incisional Negative Pressure Wound Therapy for Prevention of Postoperative Infections Following Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other); Hvidovre University Hospital (Other); Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Nana Hyldig, PhD Student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-20130010
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Surgical Wound Infection; Infection; Cesarean Section; Cesarean Section; Dehiscence; Complications; Cesarean Section; Complications; Cesarean Section, Wound, Dehiscence; Wound; Rupture, Surgery, Cesarean Section
Keywords: Randomized Controlled Trial; Economical Evaluation; Caesarean Section; postoperative wound treatment; surgical site infections; wound infections; infectious morbidity; Negative Pressure Wound Therapy; Incisional Negative Pressure Wound Therapy; Obesity
MeSH Terms: conditions — Surgical Wound Infection; Infections; Wounds and Injuries; Rupture; Wound Infection; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iNPWT (Experimental): Negative Pressure Wound Therapy (NPWT) is a mechanical wound care treatment using controlled sub-atmospheric pressure to assist and accelerate wound healing. Incisional Negative Pressure Wound Therapy (iNPWT) is a new NPWT devices, which can be used over clean closed surgical incisions. The device behaves in a similar fashion to existing conventional NPWT devices, i.e. transmission of negative pressure levels at the wound bed, tissue contraction and establishing a characteristic pattern of peri-wound blood flow and that it reduces and normalises tissue stresses at the incision
  Interventions: Device: iNPWT
- Standard wound dressing (Active Comparator): The standard postoperative wound dressing is a normal wound dressing, used over clean closed incisions.
  Interventions: Other: Standard postoperative wound dressing

INTERVENTIONS:
Device: iNPWT — The Incisional Negative Pressure Wound Therapy (iNPWT) will be applied over the clean closed incision immediately following the operation (caesarean section). In the intervention group the therapy will be left in situ for five days.
  Other Names: incisional Negative Pressure Wound Therapy
  Arms: iNPWT
Other: Standard postoperative wound dressing — A standard wound dressing will be applied over the clean closed incision immediately following the operation (caesarean section). In the control group the dressing will be left in situ for at least 24 hours as standard procedure.
  Arms: Standard wound dressing

SUMMARY:
The purpose of this study is to examine whether obese women (BMI >= 30) who give birth by caesarean section have a reduced incidence of wound infection and dehiscence when incisional Negative Pressure Wound Therapy is applied prophylactically following caesarean section.

DETAILED DESCRIPTION:
This study is a non-blinded randomised controlled trial and a concurrent Health Economic Evaluation. The study examines the effect on wound healing using incisional Negative Pressure Wound Therapy (iNPWT) compared with standard postoperative dressings in women with a BMI >= 30, who has a Caesarean Section (CS). We expect to find a lower frequency of wound complications when using iNPWT directly on primary suturing compared to standard postoperative dressings in this high-risk subpopulation.

Women, who have given informed consent, will be randomised to either intervention or control group via a computer-generated randomisation program. Elective and emergency CS will be stratified to ensure roughly equal numbers in each category of CS in each arm of the study and permit valid separate and pooled analysis. The analysis will be carried out on an intention to treat basis.

The iNPWT or standard postoperative dressings will be applied in theatre immediately following the operation. In the intervention group the therapy will be left in situ for five days corresponding to the date of removal of stitches. In the control group the dressing will be left in situ for at least 24 hours as standard procedure. Women, who do not wish to participate, will be asked for permission to use their data in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Women who can read and understand Danish
* pregestational BMI ≥ 30 kg/m2

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2013-09-10; Primary Completion 2016-10-13 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The incidence of post-CS wound infection in each study group | Within the first 30 days after surgery
  Wound infection requiring antibiotic treatment
  To be able to collect information about symptoms of infection after discharge a self-administered questionnaire will be sent to all participants within 30 days post-CS. Furthermore data on postoperative infections, recorded by diagnoses codes or surgical procedures, will be obtained from the Danish National Patient Registry

SECONDARY OUTCOMES:
Length of the primary and any secondary hospitalization | Within the first 30 days after Caesarean Section
  Primary for the health economic evaluation
Readmissions to hospital/contact to the general practitioner on suspicion of infection following caesarean section | Within the first 30 days after Caesarean Section
  Primary for the health economic evaluation
Number of Participants with a decreased health-related quality of life score as a measure of satisfaction and tolerability | Within the first 30 days after Caesarean Section
  A health-related quality of life measure, recorded in Quality Adjusted Life Years at the two interventions. The health-related quality of life score is measured 5 and 30 days post-CS. Primary for the health economic evaluation
Antibiotic treatment on suspicion of infection after Caesarean Section | Within the first 30 days after Caesarean Section
  Primary for the health economic evaluation
The cosmetic outcome as a measure of satisfaction | A 6 and 12 months follow-up
  The scar will be evaluated by a plastic surgeon at a clinical examination 6 and 12 months post-CS. After study completion pictures of the scars will be evaluated by two unbiased plastic surgeons, using two predefined scar scales.
Other wound complications after caesarean section | Within the first 30 days after Caesarean Section
  wound separation, wound exudate

CONTACTS AND LOCATIONS:
Overall Officials: Nana Hyldig, PhD Student, Study Chair — Odense University Hospital, department of Plastic Surgery, University of Southern Denmark, Faculty of Health Sciences, institute of Clinical Research, research unit, department of Gynaecology and Obstetrics
Locations (5):
- Denmark (5):
  - Aarhus University Hospital, Aarhus, Jutland
  - Hospital South West Jutland, Esbjerg, Jutland
  - Hospital Lillebaelt, Kolding Hospital, Kolding, Jutland
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No